CLINICAL TRIAL: NCT04010604
Title: A Registered Cohort Study on Spinal Muscular Atrophy
Brief Title: A Registered Cohort Study on SMA
Status: Recruiting | Type: Observational
Sponsor: Wan-Jin Chen (Other)
Responsible Party: Sponsor-Investigator, Wan-Jin Chen, The Vice-Director for the Department of Neurology, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Other Study IDs: MRCTA,ECFAHOFFMU[2019]196
Record Dates: First submitted 2019-07-01; First posted 2019-07-08 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- SMA type I
- SMA type II
- SMA type III
- Asymptomatic carriers of SMA
- Relatives of SMA patients and carriers
- Unrelated healthy controls

SUMMARY:
Spinal muscular atrophy (SMA) is an autosomal recessive disease that causes progressive muscle wasting and weakness due to loss of motor neurons in the spinal cord. This is a registered cohort of spinal muscular atrophy (SMA) type I，II and III in China. This study will provide further insights into the clinical course of SMA including overall survival, demographic characteristics, motor function, respiratory support, feeding and nutritional support, growth and development. The correlation of genotype and phenotype will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SMA types I, II and III
* Asymptomatic SMA carriers
* Relatives of SMA patients or carriers
* Unrelated healthy controls
* Participants or Parent(s)/legal guardian(s) willing and able to complete the informed consent process

Exclusion Criteria:

* Participants are unable to comply with trial procedures and visit schedule

Ages: 1 Week to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: SMA patients are diagnosed with SMN1 gene deletion or mutation.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2039-12-31 (Estimated); Study Completion 2049-12-31 (Estimated)

PRIMARY OUTCOMES:
The time to death | From date of enrollment until the date of death from any cause, assessed up to 20years
The correlation of genotype and phenotype | From date of enrollment until the date of death from any cause, assessed up to 20years
  Genotype is defined by survival motor neuron (SMN) 2 copy number(s) and phenotype is defined by clinical types and characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, First Affiliated Hospital Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No